CLINICAL TRIAL: NCT03964246
Title: Feasibility Study of Compassion Meditation Intervention for Older Veterans in Primary Care With Anxiety or Mood Disorders
Brief Title: Compassion Meditation for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E3186-P; RX003186-01 (Other Grant/Funding Number: VA Rehabilitation R&D)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Anxiety and Mood Disorders
Keywords: Feasibility Studies; Meditation, psychology
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This non-randomized feasibility study was designed to collect pilot data to establish feasibility for a future randomized controlled trial (RCT) of manualized compassion meditation (CM) group intervention for older Veterans identified through VA Primary Care clinics as having clinically significant psychological distress. The plan was to enroll 20 to 30 participants in a 10-week CM training group (with 8-10 participants in each group). As part of establishing feasibility for a subsequent large-scale RCT, the investigators also planned to enroll up to 10 additional participants in a 10-session psychoeducational group focused on topics in healthy aging. The intent for the latter was to examine the feasibility and appropriateness of employing this as a control condition in a follow-up RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Compassion Meditation (CM) intervention group (Experimental): 10-week group intervention consisting of compassion meditation training.
  Interventions: Behavioral: Compassion Meditation (CM) intervention
- Psychoeducational healthy aging group (Active Comparator): 10-week group focused on review and discussion of psychoeducational videos related to healthy aging topics
  Interventions: Other: Healthy Aging Psychoeducation

INTERVENTIONS:
Behavioral: Compassion Meditation (CM) intervention — 10 weekly 90-minute sessions. Sessions 1-3 assist participants in basic mindfulness breathing practices; sessions 4-8 focus on personal analysis of factors underlying difficulties with compassion for self or others; sessions 9 and 10 review content and assist with relapse prevention.
  [These were planned as in-person groups but due to the COVID-19 social distancing requirements that started after initiation of cohort 1, the investigators had to retool the intervention for telehealth delivery.]
  Arms: Compassion Meditation (CM) intervention group
Other: Healthy Aging Psychoeducation — The investigators planned to administer a 10-week psychoeducational in-person group focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial. This would include use of an existing library of videotaped community-focused talks, such as increasing happiness, mental resilience and health, nutrition, and physical activity.
  [Unfortunately, with the switch to telehealth format necessitated by the COVID-19 social distancing requirements, the consensus of the investigators and staff was that these proved too be too dry/"dull/academic" to be a credible attention control in a telehealth format for the target population.]
  Arms: Psychoeducational healthy aging group

SUMMARY:
Some older Veterans with psychological distress may under-utilize mental health services due to perceived stigma of symptom-focused interventions. This study was designed to examine the feasibility of a strengths-based compassion training intervention with Veterans ages > 55 years with anxiety or depressive symptoms. Although this study was focused on feasibility if successful, this line of research could open the door to a novel and effective treatment that widens acceptance by older Veterans with psychological distress.

DETAILED DESCRIPTION:
Many older Veterans in VA primary care clinics experience anxiety and depressive symptoms, but only a minority of these Veterans seek care through VA mental health services. Research suggests that some older Veterans with psychological distress under-utilize mental health services due to perceived stigma of treatments focused on mental health symptoms. However, prior research with civilians, including one study of Veterans with PTSD, suggests a strengths-focused intervention that provides group training in compassion meditation may be effective in reducing negative emotions and increasing positive emotions and well-being. This project was designed to examine the feasibility of this approach with Veterans ages > 55 years with anxiety or depression. The study was designed to guide and support development of a future larger-size, more definitive follow-up project. . If successful, this line of research could open the door to a novel and effective treatment that widens acceptance by older Veterans with psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* VA San Diego Healthcare System (VASDHS) patient
* current mild-to-moderate anxiety or depressive symptoms as defined by scores between 5 and 14 on the Patient Health Questionnaire (PHQ-9) and or Generalized Anxiety Disorders scale (GAD-7).
* stated intention to attend the 10 group sessions at the scheduled times at the VASDHS in addition to the baseline and follow-up study assessment visits, as well as to complete the outside homework assignments
* provides written informed consent for participation

Exclusion Criteria:

* no active suicidality/homicidality in the preceding six months
* untreated alcohol or substance use disorders
* changes to psychiatric medications within six months prior to the baseline evaluation
* medical and/or psychiatric instability interfering with current ability to engage in the group sessions and outside homework assignments

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton W. Palmer, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 participants enrolled (signed the ICF) and were assigned to the CM intervention, but 3 of the 25 withdrew from the study before the first intervention session. Thus 22 participants started the CM intervention (attended at least first intervention session)
Groups:
- Compassion Meditation (CM) Intervention Group: 10 weekly 90-minute sessions. Sessions 1-3 assist participants in basic mindfulness breathing practices; sessions 4-8 focus on personal analysis of factors underlying difficulties with compassion for self or others; sessions 9 and 10 review content and assist with relapse prevention.
  These were planned as in-person groups but due to the COVID-19 social distancing requirements that started after session 3 of the cohort 1, the investigators had to retool the intervention for telehealth delivery.
- Psychoeducational Healthy Aging Group: The investigators planned to examine one 10-week psychoeducational in-person group (with up to 10 participants) focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial. This would include use of an existing library of videotaped community-focused talks, such as increasing happiness, mental resilience and health, nutrition, and physical activity.
  Unfortunately, with the switch to telehealth format necessitated by the COVID-19 social distancing requirements, the consensus of the investigators and staff was that these proved too be too dry/"dull/academic" to be a credible attention control in a telehealth format for the target population.
Period: Overall Study
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Started | 22 | 0
Completed | 13 | 0
Not Completed | 9 | 0

BASELINE CHARACTERISTICS:
Population: Due to unanticipated COVID social distancing restrictions, we had to switch to a telehealth format with which the available videos for the psychoeducational sessions was too dry for a credible attention control. We began identifying more engaging videos from other sources, but with other COVID-related delays we were unable to complete this process during the study period.
  25 participants enrolled and were assigned to the CM intervention, but 3 withdrew before the first intervention session.
Groups:
- Compassion Meditation (CM) Intervention Group: Ten 90-minute group sessions: Sessions 1-3 assist participants in basic mindfulness breathing practices; sessions 4-8 focus on personal analysis of factors underlying difficulties with compassion for self or others; sessions 9 and 10 review content and assist with relapse prevention.
- Psychoeducational Healthy Aging Group: This would have been one 10-week psychoeducational in-person group (with up to 10 participants) focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial. This would include use of an existing library of videotaped community-focused talks, such as increasing happiness, mental resilience and health, nutrition, and physical activity. Unfortunately, with the switch to telehealth format necessitated by the COVID-19 social distancing requirements, the consensus of the investigators and staff was that these proved too be too dry/"dull/academic" to be a credible attention control in a telehealth form
- Total: Total of all reporting groups
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group | Total
Number analyzed (Participants) | 25 | 0 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (10.6) |  | 69.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 22 |  | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 3 |  | 3
  White | 22 |  | 22
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: The proportion of consented subjects among all screened and eligible patients.
Time Frame: 36 months
Population: Participants who were successfully contacted and verbally consented to formal telephone screening
Measure: Count of Participants; unit: Participants
Groups:
- Psychoeducational Healthy Aging Group: The investigators planned to administer a 10-week psychoeducational in-person group focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial. This would include use of an existing library of videotaped community-focused talks, such as increasing happiness, mental resilience and health, nutrition, and physical activity.
  [Unfortunately, with the switch to telehealth format necessitated by the COVID-19 social distancing requirements, the consensus of the investigators and staff was that these proved too be too dry/"dull/academic" to be a credible attention control in a telehealth format for the target population.]
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 33 | 0
Participants | 25 | 0

2. Primary Outcome: Initiation Rate
Description: The proportion of subjects who initiate the intervention among all consented subjects.
Time Frame: 4 months
Population: Participants who enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 25 | 0
Participants | 22 |

3. Primary Outcome: Completion Rate
Description: The proportion of subjects who complete 6 or more sessions (out of a total of 10 sessions) of intervention among those who start the intervention.
Time Frame: 12 weeks
Population: 22 people who attended at least the first intervention session
Measure: Count of Participants; unit: Participants
Groups:
- Compassion Meditation (CM) Intervention Group: 10-week group intervention consisting of compassion meditation training.
  Compassion Meditation (CM) intervention: 10 weekly 90-minute sessions. Sessions 1-3 assist participants in basic mindfulness breathing practices; sessions 4-8 focus on personal analysis of factors underlying difficulties with compassion for self or others; sessions 9 and 10 review content and assist with relapse prevention.
  [These were planned as in-person groups but due to the COVID-19 social distancing requirements that started after initiation of cohort 1, the investigators had to retool the intervention for telehealth delivery.]
- Psychoeducational Healthy Aging Group: 10-week group focused on review and discussion of psychoeducational videos related to healthy aging topics
  Healthy Aging Psychoeducation: The investigators planned to administer a 10-week psychoeducational in-person group focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial. This would include use of an existing library of videotaped community-focused talks, such as increasing happiness, mental resilience and health, nutrition, and physical activity.
  [Unfortunately, with the switch to telehealth format necessitated by the COVID-19 social distancing requirements, the consensus of the investigators and staff was that these proved too be too dry/"dull/academic" to be a credible attention control in a telehealth format for the target population.]
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 22 | 0
Participants | 13 |

4. Primary Outcome: Practice Time at Home
Description: Unanticipated COVID-related restrictions necessitated changing certain outcome measures. Data was not collected for this measure
Time Frame: 12 weeks
Population: Participants with data available on minutes practiced at home
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Social Connection (SCS-R) From Baseline to Post-intervention
Description: Social Connectedness Scale (SCS-R), 20-items scores, possible range = 20 to 120, higher scores reflect more connectedness
Time Frame: Baseline and 14 weeks
Population: Participants with pre- to post-intervention scores on the SCS-R
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 11 | 0
score on a scale
  Pre-intervention SCS-R total | 74.1 (14.5) |
  Post-intervention SCS-R total | 74.8 (17.1) |

6. Secondary Outcome: Mean (and SD) Change Scores for Each Inflammatory Biomarker (Hs-CRP, IL-6, and TNF- )
Description: The investigators will also examine the mean (and SD) change scores for each inflammatory biomarker (hs-CRP, IL-6, and TNF- ), as well as the association of these changes with practice time.
Time Frame: 14 weeks
Population: The COVID-19 pandemic social distancing restrictions began during the first group of participants and thus no follow-up blood samples could be collected for this or subsequent groups. Due to absence of follow-up blood draws for the initial group and an absence of baseline and follow-up data for the remaining participants, the inflammatory biomarker outcomes could not be examined.
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Depression and Anxiety From Baseline to Post-intervention
Description: Brief Symptom Inventory-18 (BSI; depression, anxiety, and somatization) Global Severity Index (GSI). Each of the 18 items range from a score of 0-4; total score ranges from 0-72 with higher scores indicating worse function.
Time Frame: Baseline and 14 weeks
Population: Participants with pre- and post-intervention data for BSI-GSI
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 10 | 0
score on a scale
  Pre-Intervention BSI- GSI | 17.9 (12.0) |
  Post-Intervention BSI-GSI | 14.9 (10.4) |

8. Secondary Outcome: Satisfaction With Life (SWLS) From Baseline to Post-intervention
Description: Satisfaction With Life Scale (SWLS); 5-items, range 5 to 35, higher scores represent greater satisfaction
Time Frame: Baseline and 14 weeks
Population: Participants with pre-post scores on the SWLS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 10 | 0
score on a scale
  Pre-Intervention SWLS total | 18.0 (9.7) |
  Post-Intervention SWLS total | 21.0 (8.8) |

9. Secondary Outcome: Change in Positive Emotions (mDES) From Baseline to Post-intervention
Description: 10-item positive emotions subscale of the 20-item modified Differential Emotions Scale (mDES); scores on this subscale have a potential range of 0 to 40 with higher scores reflecting more positive emotions.
Time Frame: Baseline and 14 weeks
Population: Participants with pre- and post-intervention scores on the mDES positive emotions subscale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
Number analyzed (Participants) | 11 | 0
score on a scale
  Pre-Intervention mDES Positive Emotions subscale total | 21.7 (7.8) |
  Post-Intervention mDES Positive Emotions subscale total | 21.0 (7.8) |

ADVERSE EVENTS:
Time Frame: 12 weeks (baseline evaluation to final study visit)
Description: Clinicaltrials.gov definitions are used.
Groups:
- Psychoeducational Healthy Aging Group: This would have been one 10-week psychoeducational in-person group (with up to 10 participants) focused on topics in healthy aging to examine its feasibility as a control condition for a subsequent randomized controlled trial.
Arm/Group | Compassion Meditation (CM) Intervention Group | Psychoeducational Healthy Aging Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/0

LIMITATIONS AND CAVEATS:
Unanticipated COVID-related social distancing restrictions necessitated changing to remote assessment and intervention during the first intervention cohort and throughout the remainder of the trial. The lessons learned are valuable in the context of this as a feasibility study, could potentially help future studies of the intervention focused on Veterans with transportation or geographic distance limitations, but hindered our completion of some of the originally planned components of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT03964246/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT03964246/ICF_002.pdf